CLINICAL TRIAL: NCT01656902
Title: A Prospective Randomized Controlled Multicenter Phase-III Clinical Study to Evaluate the Safety and Effectiveness of NOVOCART® 3D Plus Compared to the Standard Procedure Microfracture in the Treatment of Articular Cartilage Defects of the Knee
Brief Title: Phase III Study to Evaluate Safety and Effectiveness of NOVOCART 3D Plus vs. Microfracture in Knee Cartilage Defects
Acronym: N3D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tetec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-1202
Record Dates: First submitted 2012-07-20; First posted 2012-08-03 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2021-10

CONDITIONS: Traumatic Articular Cartilage Defects in the Knee Joint
Keywords: Autologous Chondrocyte Transplantation; NOVOCART 3D plus; knee joint pain; safety; efficacy; treatment; TETEC; cartilage; ACT; cartilage repair; tissue; MOCART
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N3D plus (Experimental): NOVOCART® 3D plus (Autologous Chondrocyte Transplantation System)
  Interventions: Drug: NOVOCART® 3D plus
- Microfracture (Active Comparator): Microfracture is the standard care surgery.
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Drug: NOVOCART® 3D plus — Two-Step intervention: 1) cartilage cells are collected from the patient during arthroscopy 2) collected cartilage cells are cultivated in a sterile environment, seeded in an organic matrix scaffold and implanted into the defect location (knee, femur)
  Other Names: Matrix-associated autologous chondrocyte implantation
  Arms: N3D plus
Procedure: Microfracture — single-step treatment: defect location (knee, femur) is debrided, then bone plate is drilled mechanically to allow cells from the bone marrow to move to the defect location and to develop a scar tissue
  Other Names: Microfracture according to Steadman
  Arms: Microfracture

SUMMARY:
In this phase 3 clinical trial, a second generation ACI (autologous chondrocyte implantation technique) is compared to standard of care therapy (microfracture) to treat traumatic cartilage defects of the knee for efficacy and safety. The investigated study treatment NOVOCART 3D plus is a biphasic biological scaffold which contains cultivated chondrocytes derived from the patient in a previous tissue harvest procedure. Allocation to the study treatment is done by randomization in a ration of 2:1 in favor to ACI (investigational product). Follow-up data for efficacy is collected for 2 years: follow-up visits are performed 6 weeks, 3 months, 6 months, 12 months, 18 months and 24 months after treatment; additional data for safety will be collected for up to 5 years: 36, 48, and 60 months after treatment. The study involves knee surgery (by arthroscopy, or mini-arthrotomically for implantation surgery), and blood withdrawal for safety within the first year after treatment. Initial imaging is required at baseline. Optional MRI imaging and biomarker collection is done as substudy at specific sites only.

DETAILED DESCRIPTION:
For the cartilage cell product NOVOCART® 3D plus, which is used in the study described here, the company TETEC AG obtained an expanded production authorization from the medication monitoring authorities in compliance with Section 13, Para. 1 of the Medicinal Products Act in 2003. This entitles TETEC AG to produce the pharmaceutical product and already distribute it. More than 6000 patients were already successfully treated with NOVOCART® 3D in Europe since 2003. In order to obtain a general market authorization for NOVOCART® 3D plus, this control group study is conducted, in which the superiority of the safety and effectiveness of carrier-bound Autologous Chondrocyte Transplantation with NOVOCART® 3D plus compared to the standard of care microfracture surgery needs to be proven. This study further aims at developing and validating known and new biologic markers for the quality and clinical efficacy of the product as requested in the context of identity, purity and potency characteristics of the medicinal/investigational product.

The patients will receive one of the therapeutic procedures in the study. The treatment procedure which will be used will be decided by a previously specified randomization process. This type of study meets the high quality requirements of the statutorily specified safety and quality regulations which are also referred to as "Good Clinical Practice" (GCP). The probability of the patient being allocated to one of the two treatments is 2:1; that is, an approx. 67% probability of therapy with NOVOCART® 3D plus and an approx. 33% probability of therapy with microfracture. Neither the patient, nor the investigator will be able to influence the treatment assignment.

Patients will be screened for eligibility at the Screening Visit. Each patient will remain in the study for 24 months post-implant for the effectiveness assessments, and then an additional three years to complete the planned post-market phase. Each patient will be in the study for up to five years.

Cells and tissues collected from this study will be used in other in vitro-controlled experiments aimed at developing and validating known and novel biologic markers to quantify cell quality in the context of identity, purity and potency. Prognostic values of these biologic markers will be examined by correlating them with clinical data collected in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 65 years old at screening OR (in selected countries only) is a pediatric patient (14-17 years old) with closed epiphyseal growth plate (confirmation of closure of epiphyseal growth plate of the index knee by x-ray or MRI required).
2. Patient has a localized articular cartilage defect of the femoral condyle or the trochlea of the knee. 2 localized cartilage defects are accepted if the total defect size is ≤ 6 cm2 and the size of each individual lesion is ≥ 2 cm2, both cartilage defects are located at the femoral condyle and/or the trochlea and both cartilage defects are to be treated with NOVOCART 3D plus or microfracture.
3. Patient has a defect size is between 2 and 6 cm2. Note: defect size can be estimated by MRI at visit 1 if no data is available from medical history.
4. Patient has an intact articulating joint surface (not higher than Grade 2 International Cartilage Repair Society classification, no kissing lesions). Note: ICRS classification can be estimated by MRI at visit 1 if no data is available from medical history.
5. Patient has an intact meniscus; a maximum of 50% resection is allowed. Note: status of meniscus can be estimated at visit 1 if no data is available from medical history.
6. Patient has a stable knee joint or sufficiently reconstructed ligaments. If not, ligament repair must be done before, during or within 6 weeks after cartilage treatment (ACT/microfracture).
7. Patient has free range of motion of the affected knee joint or ≤ 10° of extension and flexion loss.
8. Patient has a defect-grade of III or IV according to the ICRS classification. Note: ICRS classification can be estimated by MRI at visit 1 if not data is available from medical history.
9. Patient has a baseline score of 60/100 on the 2000 International Knee Documentation Committee (IKDC) subjective knee evaluation.
10. Patient is willing and able to give written informed consent to participate in the study and to comply with all study requirements, including attending all follow-up visits and assessments and postoperative rehabilitation regimen.
11. Mandatory for France only: Patient benefits of a health insurance regimen.

Exclusion Criteria (pre-operative):

1. Patient is the investigator or any subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.
2. Patient is unable to undergo magnetic resonance imaging (MRI).
3. Patient has prior surgical treatment of the target knee using mosaicplasty, autologous chondrocyte transplantation and/or microfracture. Note: prior diagnostic arthroscopies with debridement and lavage are acceptable. Ligament repair is accepted, if performed before, during or within 6 weeks after cartilage treatment (ACT/microfracture).
4. Patient has radiologically apparent degenerative joint disease in the target knee as determined by Kellgren and Lawrence grade > 2 (see Appendix A).
5. Patient has chronic inflammatory arthritis and/or infectious arthritis.
6. Patient has joint space narrowing > 1/3 in the target knee when compared to the other knee or smaller than 3 mm joint space measured on x-ray.
7. Patient has malalignment (valgus- or varus-deformity) in the target knee. Note: In suspected cases, the mechanical axis must be established radiographically by complete leg imaging in standing position and in a.p. or rather p.a. projection. The Mikulicz line is not allowed to deviate more than 5 mm of the eminentia intercondylaris. If alignment is necessary, surgery has to be performed before, during or within 6 weeks after cartilage treatment (ACT/microfracture).
8. Patient has prior surgical treatment of clinical relevance of the target knee.
9. Patient has an osteochondral defect.
10. Patient has bilateral lower limb pain or low back pain.
11. Patient has a known systemic connective tissue disease.
12. Patient has a current uncontrolled diabetes.
13. Patient has a known history of autoimmune disease.
14. Patient has a known history of immunological suppressive disorder or is taking immunosuppressants.
15. Patient is currently systemically or intra-articularly taking steroids and/or has used steroids within the last 30 days prior to screening visit 1.
16. The patient has a history of HIV/AIDS.
17. The patient has a history of syphilis (Treponema pallidum).
18. The patient has an active hepatitis B or C infection with verified antigens. Note: Patients with a cured hepatitis B or C infection and/or verified antibodies are not excluded.
19. The patient has at the site of surgery an active systemic or local microbial infection, eczematization or inflammable skin alterations (including protozoonosis: Babesiosis, Trypanosomiasis (e.g. Chagas-Disease), Leishmaniasis, persistent bacterial infections, like Brucellosis, spotted and typhus fever, other Rickettsiosis, Leprosy, Recurrent Fever, Melioidosis or Tularaemia).
20. Patient has a known history of cancer within the past 5 years.
21. Patient has a known history of osteoporosis; also patients with primary hyperparathyroidism or hyperthyroidism without satisfactory treatment, chronic renal failure or patients with prior pathological fractures independent of the genesis are excluded.
22. Patient has any degenerative muscular or neurological condition that would interfere with evaluation of outcome measures including but not limited to Parkinson's disease, amyotrophic lateral sclerosis (ALS), or multiple sclerosis (MS).
23. Patient has a body mass index (BMI) higher than 35 kg/m2.
24. Patient is a woman who is pregnant or lactating. Note: contraception is indicated for female patients of childbearing potential until the day of cartilage treatment. Female patients who are unwilling to practice a medically acceptable method of birth control until the day of cartilage treatment cannot be included.
25. Patient is currently participating, or has participated in any other clinical study within 3 months prior to the screening visit.
26. Patient has known current or recent history of illicit drug or alcohol abuse or dependence
27. Patient has psychiatric or cognitive impairment that, in the opinion of the investigator, would interfere with the patient's ability to comply with the study requirements, e.g., Alzheimer's disease.
28. Patient has any other condition, which, in the opinion of the investigator, would make the patient unsuitable for the study.
29. Patient has a history of HTLV.

Intra-operative Inclusion Criteria:

1. Patient is not pregnant as confirmed by urine pregnancy test before arthroscopy.
2. Patient has a localized articular cartilage defect of the femoral condyle or the trochlea of the knee. 2 localized cartilage defects are accepted if the total defect size is up to 6 cm2 and the size of each individual lesion is at least 2 cm2, both cartilage defects are located at the femoral condyle and/or the trochlea and both cartilage defects are to be treated with NOVOCART 3D plus or microfracture.
3. Patient has a defect size of 2 to 6 cm2 post-debridement.
4. Patient has an intact articulating joint surface (at least (or higher) Grade 2 International Cartilage Repair Society classification) no kissing lesions).
5. Patient has an intact meniscus; a maximum of 50% resection is allowed (no indication for concurrent meniscus transplant).
6. Patient has a stable knee joint or sufficiently reconstructed ligaments. If not, ligament repair must be done during or within 6 weeks after cartilage treatment (ACT/microfracture).
7. Patient has a defect grade of III or IV according to the ICRS classification.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Subjective IKDC score | Baseline assessment to 24-month follow-up assessment
  The primary endpoint is the change from baseline in the "2000 International Knee Documentation Committee" (IKDC) subjective score to 24-month visit.
  The IKDC will be recorded for NOVOCART® 3D plus and microfracture patients at baseline visit 1 and at the 6 weeks, 3-, 6-, 12-, 24-, 36-, 48,- and 60-month follow-up assessments.

SECONDARY OUTCOMES:
IKDC objective physician score | Baseline assessment to 24-month follow-up assessment
  The IKDC objective physician score will be recorded for both arms at baseline visit 1 and at the 6 weeks, 3-, 6-, 12-, 24-, 36-, 48,- and 60-month follow-up assessments. A sequentially rejecting, hierarchical test procedure will be employed to test these secondary endpoints in the a-priori defined order given here after the test primary efficacy variable was passed.
  The change from baseline to the 24-month visit in the IKDC objective physician score and from baseline to the 24-month visit will be evaluated.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline assessment to 24-month follow-up assessment
  The KOOS will be recorded for both arms at baseline visit 1 and at the 6 weeks, 3-, 6-, 12-, 24-, 36-, 48,- and 60-month follow-up assessments.
  A sequentially rejecting, hierarchical test procedure will be employed to test these secondary endpoints in the a-priori defined order given here after the test primary efficacy variable was passed. The change from baseline to 24-month visit in the Knee Injury and Osteoarthritis Outcome Score (KOOS) and from baseline to 24-month visit will be evaluated.
MOCART Score (MRI) | Baseline assessment to the 24-month assessment
  Another secondary efficacy endpoint is the in vivo performance (grading on quality of cartilage fill) measured by the change from baseline to the 36-month assessment of the Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score. These assessments will be performed on a subset of patients (64 in NOVOCART and 32 in microfracture arm).
  The MRI will be recorded at 3, 12, 24 and 60 months follow-up visit.
Health-related quality of life as measured by the SF-36 survey | Baseline assessment to 24-month follow-up assessment
  Another secondary efficacy endpoint is the change from baseline to the 24-month visit in the SF-36 to measure clinical utility and summarize health-related quality-of-life and cost-effectiveness. The SF-36 will be recorded for NOVOCART® 3D plus and microfracture patients at baseline visit 1 and at the 6 weeks, 3-, 6-, 12-, 24-, 36-, 48,- and 60-month follow-up assessments.
Surgical time (cut-to-suture time) | Transplantation (24 +-5 days post-arthroscopy) and/or arthroscopy (>= 1 day after screening), depending on the study arm
  The surgical time will be measured in minutes and recorded for NOVOCART® 3D plus patients at arthroscopy (>= 1 day after screening) and transplantation (24 +-5 days post-arthroscopy); for microfracture patients surgical time will be measured in minutes and recorded at arthroscopy (>= 1 day after screening).
Length of incision | Only for verum group at transplantation (24 +-5 days post-arthroscopy)
  The length of incision will be measured in cm and recorded for NOVOCART® 3D plus patients at transplantation (24 +-5 days post-arthroscopy)
Any unanticipated adverse event | Baseline assessment up to 60-months follow-up assessment
  Event descriptions, onset, resolution dates, relationship to the IP and procedures of any AEs will be recorded. Each event will be categorized by seriousness and intensity to facilitate complete safety reporting throughout the trial.
  While comparisons between treatment groups can be made for each class of AE, there is no statistical hypothesis governing acceptance of this endpoint at the end of the clinical study because of the different AE profiles associated with the two treatment arms.
Treatment Failure | From completion of study treatment until 60-months follow-up assessment
  Any event related to a diagnosed failure of the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Angele, Prof., Principal Investigator — Universitätsklinikum Regensburg
Locations (35):
- Privatklinik Doebling, Vienna, Austria
- Czechia (7):
  - Fakultni nemocnice Brno - Ortopedicka klinika, Brno
  - Urazova nemocnice v Brne - Traumatologie, Brno
  - NH Hospital, a.s., Ortopedicke oddeleni nemocnice Horovice, Hořovice
  - Fakultni nemocnice Hradec Kralove - Ortopedicka klinika, Hradec Králové
  - Pardubicka nemocnice, Pardubice
  - Fakultni nemocnice v Motole, Prague
  - UVN - Vojenska fakultni nemocnice Praha, Prague
- France (4):
  - Hôpital Ambroise Paré - Service de Chirurgie Orthopedique et Traumatologie, Boulogne-Billancourt
  - Polyclinique Saint-Roch, Montpellier
  - Clinique V - Clinique du Sport, Paris
  - CHU de Saint-Etienne Hôpital Nord - Service orthopedie et traumatologie, Saint-Priest-en-Jarez
- Germany (4):
  - Universitaetsklinikum Freiburg - Klinik fuer Orthopaedie, Freiburg im Breisgau
  - Theresienkrankenhaus, Mannheim
  - Orthopädische Klinik und Poliklinik der LMU München, München
  - Universitätsklinikum Regensburg, Regensburg
- Hungary (5):
  - Uzsoki utcai Kórház, Budapest
  - Petz Aladár Megyei Oktató Kórház, Győr
  - B-A-Z Megyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
  - Markusovszky Egyetemi Oktatókórház, Szombathely
  - Kastélypark Klinika, Tata
- Latvia (2):
  - Hospital of Traumatology and Orthopaedics, Trauma Department, Riga
  - Orto Clinic, Riga
- Lithuania (5):
  - Kaunas clinical hospital, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda university hospital, Klaipėda
  - JSC "Kardiolita", Vilnius
  - JSC "SK Impeks Medicinos Diagnostikos Centras", Vilnius
- Poland (5):
  - Szpital sw. Lukasza BGL Sp z o.o. S.K.A., Bielsko-Biala
  - Samozdzielny Publiczny Zaklad Opieki Zdrowotnej Miejskiego Szpitala Zespolonego, Częstochowa
  - Szpital Angelius, Katowice
  - Samozdzielny Publiczny Wojewodzki Szpital Chirurgii Urazowej, Piekary Śląskie
  - Centrum Medycyny Sportowej, Warsaw
- Universitätsklinikum Basel, Basel, Switzerland
- Royal Devon and Exeter Hospital, Exeter, United Kingdom